CLINICAL TRIAL: NCT02496208
Title: A Phase 1 Study of Cabozantinib Plus Nivolumab (CaboNivo) Alone or in Combination With Ipilimumab (CaboNivoIpi) in Patients With Advanced/Metastatic Urothelial Carcinoma and Other Genitourinary Tumors
Brief Title: Cabozantinib S-malate and Nivolumab With or Without Ipilimumab in Treating Patients With Metastatic Genitourinary Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-02379; NCI-2014-02379 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 15-C-0160; 150160; P141706; 9681 (Other: National Cancer Institute LAO); 9681 (Other: CTEP); UM1CA186712 (NIH); UM1CA186716 (NIH); UM1CA186717 (NIH); ZIABC011078 (NIH)
Record Dates: First submitted 2015-07-08; First posted 2015-07-14 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Bladder Small Cell Neuroendocrine Carcinoma; Bladder Squamous Cell Carcinoma; Bladder Urothelial Carcinoma; Clear Cell Renal Cell Carcinoma; Invasive Bladder Plasmacytoid Urothelial Carcinoma; Invasive Bladder Sarcomatoid Urothelial Carcinoma; Invasive Sarcomatoid Urothelial Carcinoma; Kidney Medullary Carcinoma; Malignant Genitourinary System Neoplasm; Malignant Solid Neoplasm; Penile Carcinoma; Penile Squamous Cell Carcinoma; Renal Cell Carcinoma; Renal Pelvis Urothelial Carcinoma; Sarcomatoid Renal Cell Carcinoma; Stage III Bladder Cancer AJCC v8; Stage III Penile Cancer AJCC v8; Stage III Renal Cell Cancer AJCC v8; Stage III Renal Pelvis and Ureter Cancer AJCC v8; Stage III Renal Pelvis Cancer AJCC v8; Stage III Ureter Cancer AJCC v8; Stage III Urethral Cancer AJCC v8; Stage IV Bladder Cancer AJCC v8; Stage IV Penile Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v8; Stage IV Renal Pelvis and Ureter Cancer AJCC v8; Stage IV Ureter Cancer AJCC v8; Stage IV Urethral Cancer AJCC v8; Ureter Urothelial Carcinoma; Urethral Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Urogenital Neoplasms; Penile Neoplasms; Urinary Bladder Neoplasms; Ureteral Neoplasms; Urethral Neoplasms | interventions — Biopsy; Specimen Handling; cabozantinib; Ipilimumab; CTLA-4 Antigen; Magnetic Resonance Spectroscopy; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part I (cabozantinib s-malate, nivolumab) (Experimental): Patients receive cabozantinib s-malate PO QD on days 1-28 and nivolumab IV over 30 minutes on days 1 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. After 21 cycles, patients receive nivolumab IV over 30 minutes every 4 weeks in the absence of disease progression or unacceptable toxicity. After progression, patients may receive cabozantinib s-malate PO, nivolumab IV, and ipilimumab IV at the part II RP2D for 4 cycles followed by cabozantinib s-malate PO QD and nivolumab IV every 2 weeks or 4 weeks if post-cycle 21 in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography or magnetic resonance imaging and collection of blood samples throughout the trial. Patients may also undergo echocardiography at baseline and biopsies throughout the trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Cabozantinib S-malate; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab
- Part II (cabozantinib s-malate, nivolumab, ipilimumab) (Experimental): See detailed description.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Cabozantinib S-malate; Procedure: Computed Tomography; Procedure: Echocardiography Test; Biological: Ipilimumab; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsies
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cabozantinib S-malate — Given PO
  Other Names: BMS-907351; Cabometyx; Cometriq; XL 184; XL-184; XL184
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo echocardiography
  Other Names: EC; Echocardiography
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
  Arms: Part II (cabozantinib s-malate, nivolumab, ipilimumab)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo

SUMMARY:
This phase I trial studies the side effects and best doses of cabozantinib s-malate and nivolumab with or without ipilimumab in treating patients with genitourinary (genital and urinary organ) tumors that have spread from where it first started (primary site) to other places in the body (metastatic). Cabozantinib s-malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as nivolumab and ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. It is not yet known whether giving cabozantinib s-malate and nivolumab alone or with ipilimumab works better in treating patients with genitourinary tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the dose limiting toxicity (DLT) and recommended phase II dose (RP2D) of the combination of cabozantinib s-malate (cabozantinib) and nivolumab (cabo-nivo) and separately the combination of cabozantinib, nivolumab and ipilimumab (cabo-nivo-ipi) in patients with genitourinary tumors. (Phase I) II. Assess safety and tolerability of cabozantinib, nivolumab and ipilimumab (cabo-nivo-ipi) in patients with genitourinary tumors at this novel dose. (Dose Level 8 Cohort)

SECONDARY OBJECTIVES:

I. Preliminarily evaluate the activity, as determined by objective response rate using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and the modified Immune-Related Response Criteria (irRC), derived from RECIST 1.1, of:

Ia. Cabo-nivo and cabo-nivo-ipi in patients with advanced/refractory metastatic urothelial carcinoma (checkpoint inhibition therapy naive) and with renal cell carcinoma in the second-line and beyond setting.

Ib. Cabo-nivo in patients with adenocarcinoma and with rare histologies (including squamous or small cell carcinomas of the bladder, renal medullary carcinoma, sarcomatoid bladder and renal cell carcinomas, plasmacytoid carcinoma of the bladder and others) in the first line or beyond setting.

Ic. Cabo-nivo in patients with urothelial carcinoma previously treated with checkpoint inhibition therapy in the second line or beyond setting.

Id. Cabo-nivo-ipi in patients with squamous cell carcinoma of the penis.

II. To evaluate the activity as determined by progression free survival (PFS) and overall survival (OS) of:

IIa. Cabo-nivo and cabo-nivo-ipi in patients with advanced/refractory metastatic urothelial carcinoma (checkpoint inhibition therapy naive) or with renal cell carcinoma in the second-line and beyond setting.

IIb. Cabo-nivo in patients with adenocarcinoma and with rare histologies (including squamous, small cell carcinomas of the bladder, renal medullary carcinoma, sarcomatoid bladder and renal cell carcinomas, plasmacytoid carcinoma of the bladder and others) in the first line or beyond setting.

IIc. Cabo-nivo in patients with urothelial carcinoma previously treated with checkpoint inhibition therapy in the second line or beyond setting.

IId. Cabo-nivo-ipi in patients with squamous cell carcinoma of the penis. III. To obtain additional data to evaluate the safety of both combinations in patients with clear cell renal cell carcinoma (ccRCC).

IV. To assess the number of malignant soft tissue and bone lesions on fludeoxyglucose F-18 (18F-FDG) positron emission tomography (PET)/computed tomography (CT) (scan 1) versus combined fluorine F 18 sodium fluoride (18F-NaF) and 18F-FDG PET/CT (scan 2).

V. To assess response assessment by RECIST 1.1 using CT of the chest, abdomen, and pelvis with intravenous (IV) contrast versus assessment by combined 18F-NaF and 18F-FDG PET/CT (scan 2) using number of malignant and change (modified PET RECIST [PERCIST]) of soft tissue and bone lesions.

VI. To test the feasibility of automated density and volume application (ADaVA) as a means of assessing tumor response.

VII. To assess PDL-1 and MET expression data and in exploratory fashion analyze their association to response or clinical benefit.

EXPLORATORY OBJECTIVES:

I. To assess overall response rates (ORR) on patients who have been challenged or re-challenged with ipilimumab therapy post disease progression.

II. To assess effects of treatment in patients with bone-only disease. III. To use circulating tumor deoxyribonucleic acid (ctDNA) analysis to assess the level of ctDNA at multiple time points during therapy and correlate with outcomes (e.g., objective responses, disease burden, PFS, OS, and adverse events).

OUTLINE: This is a dose-escalation study. Patients are assigned to 1 of 2 treatment arms.

PART I: Patients receive cabozantinib s-malate orally (PO) once daily (QD) on days 1-28 and nivolumab intravenously (IV) over 30 minutes on days 1 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. After 21 cycles, patients receive nivolumab IV over 30 minutes every 4 weeks in the absence of disease progression or unacceptable toxicity. After progression, patients may receive cabozantinib s-malate PO, nivolumab IV, and ipilimumab IV at the part II RP2D for 4 cycles followed by cabozantinib s-malate PO QD and nivolumab IV every 2 weeks or 4 weeks if post-cycle 21 in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography or magnetic resonance imaging and collection of blood samples throughout the trial. Patients may also undergo echocardiography at baseline and biopsies throughout the trial.

PART II: Patients receive cabozantinib s-malate PO QD on days 1-21, nivolumab IV over 30 minutes on day 1, and ipilimumab IV over 90 minutes on day 1 of each cycle. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. After completion of 4 cycles with ipilimumab, patients continue receiving cabozantinib s-malate PO QD on days 1-28 and nivolumab IV over 30 minutes on days 1 and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. After 21 cycles, patients receive nivolumab IV over 30 minutes every 4 weeks in the absence of disease progression or unacceptable toxicity. After progression, patients may receive cabozantinib s-malate PO, nivolumab IV, and ipilimumab IV at the part II RP2D for 4 cycles followed by cabozantinib s-malate PO QD and nivolumab IV every 2 weeks or 4 weeks if post-cycle 21 in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography or magnetic resonance imaging and collection of blood samples throughout the trial. Patients may also undergo echocardiography at baseline and biopsies throughout the trial.

After completion of study treatment, patients are followed up at 16 weeks, and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the phase I portion must have:

  * Histologically confirmed diagnosis of metastatic, genitourinary solid tumor
  * Metastatic disease defined as new or progressive lesions on cross-sectional imaging; patients must have at least:

    * One evaluable site of disease
    * Or, appearance of one new bone lesion
* Patients in the expansion portion must have:

  * Histologically confirmed diagnosis of metastatic:

    * Urothelial carcinoma of the bladder, urethra, ureter, renal pelvis, OR
    * Clear cell renal cell carcinoma OR
    * Adenocarcinoma of the bladder OR
    * Non-resectable squamous cell carcinoma of the penis OR
    * Squamous or small cell carcinoma of the bladder, renal medullary carcinoma (RMC), sarcomatoid bladder and renal cell carcinomas, plasmacytoid carcinoma of the bladder or other rare bladder/kidney cancer histology AND
  * Patients with urothelial cancer or renal cell carcinoma must have progressive metastatic disease defined as new or progressive lesions on cross-sectional imaging; patients must have at least:

    * One measurable site of disease (according to RECIST criteria) or bone disease by NaF PET/CT
* Patients must have either progressed on at least one standard therapy or there must be no standard treatment that has been shown to prolong survival for the patient's disease (patients with urothelial carcinoma who are cisplatin-ineligible may receive protocol therapy as a first line therapy); patients may have received any number of prior cytotoxic agents
* Age >= 18 years on day of consent. Because no dosing or adverse event data are currently available on the use of cabozantinib in combination with nivolumab and ipilimumab in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* Karnofsky performance status >= 70%
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,200/mcL
* Platelets >= 75,000/mcL
* Total bilirubin =< 1.5 x upper limit of normal (ULN); for subjects with known Gilbert's disease or similar syndrome with slow conjugation of bilirubin, total bilirubin =< 3.0 mg/dL
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 x institutional upper limit of normal (ULN)
* Creatinine =< 1.5 x ULN OR creatinine clearance >= 40 mL/min/1.73 m^2 (calculated using the Chronic Kidney Disease-Epidemiology Collaboration [CKD-EPI] equation or Cockcroft-Gault formula) for patients with creatinine levels above institutional normal
* Hemoglobin >= 9 g/dL
* Serum albumin >= 2.8 g/dL
* Lipase and amylase =< 2.0 x ULN and no radiologic or clinical evidence of pancreatitis
* Urine protein/creatinine ratio (UPCR) =< 2
* Serum phosphorus >= lower limit of normal (LLN) (if below LLN, for asymptomatic patients replacement may be initiated if clinically indicated without delaying the start of study treatment)
* Serum calcium >= LLN (if below LLN, for asymptomatic patients replacement may be initiated if clinically indicated without delaying the start of study treatment)
* Serum magnesium >= LLN (if below LLN, for asymptomatic patients replacement may be initiated if clinically indicated without delaying the start of study treatment)
* Serum potassium >= LLN (if below LLN, for asymptomatic patients replacement may be initiated if clinically indicated without delaying the start of study treatment)
* Women of childbearing potential must have a negative pregnancy test at screening; women of childbearing potential include women who have experienced menarche and who have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are not postmenopausal; postmenopause is defined as amenorrhea >= 12 consecutive months; Note: women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, ovarian suppression or any other reversible reason
* The effects of the drugs used in this trial on the developing human fetus are unknown; however, cabozantinib was embryolethal in rats at exposures below the 140 mg dose in the label, with increased incidences of skeletal variations in rats and visceral variations and malformations in rabbits; for this reason and because tyrosine kinase inhibitors agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception, as defined below, prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and for 7 months after completion of all study medications; women treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and for 5 months after completion of all study medications
* Sexually active subjects (men and women) must agree to use medically accepted barrier methods of contraception (e.g., male or female condom) during the course of the study and for 5 or 7 months for women or men respectively, after the last dose of study drugs, even if oral contraceptives are also used; all subjects of reproductive potential must agree to use both a barrier method and a second method of birth control during the course of the study and for 5 or 7 months for women and men respectively after the last dose of study drugs
* Tissue availability for PD-L1 expression is mandatory for enrollment; however if archived tissue is unavailable the patient will be given the option to consent to pre and post treatment tissue biopsies; tissue biopsies will be collected pretreatment (prior to the first dose of therapy) and post treatment (after at least 1 dose, preferably 2 doses of nivolumab)
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* The subject has received cytotoxic chemotherapy (including investigational cytotoxic chemotherapy) or biologic agents (e.g., cytokines or antibodies) within 3 weeks, or nitrosoureas/mitomycin C within 6 weeks before the first dose of study treatment
* Patients who have been previously treated with MET or VEGFR inhibitors (except for patients on renal cell cancer [RCC] cohort) are not eligible for the expansion cohorts but can enroll in the phase I portion
* Prior treatment with any therapy on the PD-1/PD-L1 axis or CTLA-4 inhibitors unless enrolling the urothelial carcinoma with previous checkpoint inhibition therapy expansion cohort
* The subject has received radiation therapy:

  * To the thoracic cavity or abdomen within 3 months before the first dose of study treatment, or has ongoing complications, or is without complete recovery and healing from prior radiation therapy
  * To bone or brain metastasis within 3 weeks before the first dose of study treatment
  * To any other site(s) within 28 days before the first dose of study treatment
* The subject has received radionuclide treatment within 6 weeks of the first dose of study treatment
* The subject has received prior treatment with a small molecule kinase inhibitor within 14 days or five half-lives of the compound or active metabolites, whichever is longer, before the first dose of study treatment
* The subject has received prior treatment with hormonal therapy within 14 days or five half-lives of the compound or active metabolites, whichever is longer, before the first dose of study treatment; subjects receiving gonadotropin-releasing hormone (GnRH) agonists and antagonists are allowed to participate
* The subject has received any other type of investigational agent within 28 days before the first dose of study treatment
* The subject has not recovered to baseline or Common Terminology Criteria for Adverse Events (CTCAE) =< grade 1 from toxicity due to all prior therapies except alopecia and other non-clinically significant adverse events (AEs) defined as lab elevation with no associated symptoms or sequelae
* The subject has active brain metastases or epidural disease; subjects with brain metastases previously treated with whole brain radiation or radiosurgery or subjects with epidural disease previously treated with radiation or surgery who are asymptomatic and do not require steroid treatment for at least 2 weeks before starting study treatment are eligible; neurosurgical resection of brain metastases or brain biopsy is permitted if completed at least 3 months before starting study treatment; baseline brain imaging with contrast-enhanced CT or magnetic resonance imaging (MRI) scans for subjects with known brain metastases is required to confirm eligibility
* The subject has prothrombin time (PT)/international normalized ratio (INR) or partial thromboplastin time (PTT) test >= 1.5 x the laboratory ULN within 7 days before the first dose of study treatment
* No concomitant treatment with warfarin is permitted. Aspirin (up to 325 mg/day), thrombin or factor Xa inhibitors, low-dose warfarin (=<1 mg/day), prophylactic and therapeutic low molecular weight heparin (LMWH) are permitted
* The subject requires chronic concomitant treatment of strong CYP3A4 inducers (e.g., dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital, and St. John's wort); Because the lists of these agents are constantly changing, it is important to regularly consult medical reference texts such as the Physicians' Desk Reference may also provide this information; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* The subject has experienced any of the following:

  * Clinically-significant gastrointestinal bleeding within 6 months before the first dose of study treatment
  * Hemoptysis of >= 0.5 teaspoon (2.5 mL) of red blood within 3 months before the first dose of study treatment
  * Any other signs indicative of pulmonary hemorrhage within 3 months before the first dose of study treatment
* The subject has tumor invading any major blood vessels
* The subject has evidence of tumor invading the gastrointestinal (GI) tract (esophagus, stomach, small or large bowel, rectum or anus), or any evidence of endotracheal or endobronchial tumor within 28 days before the first dose of cabozantinib
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:
* Cardiovascular disorders including:

  * Congestive heart failure (CHF): New York Heart Association (NYHA) class III (moderate) or class IV (severe) at the time of screening
  * Concurrent uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mmHg systolic, or > 90 mmHg diastolic despite optimal antihypertensive treatment within 7 days of the first dose of study treatment
  * The subject has a corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms within 28 days before randomization; Note: if initial QTcF is found to be > 500 ms, two additional electrocardiograms (EKGs) separated by at least 3 minutes should be performed; if the average of these three consecutive results for QTcF is =< 500 ms, the subject meets eligibility in this regard
  * Any history of congenital long QT syndrome
  * Any of the following within 6 months before the first dose of study treatment:

    * Unstable angina pectoris
    * Clinically-significant cardiac arrhythmias
    * Stroke (including transient ischemic attack [TIA], or other ischemic event)
    * Myocardial infarction
    * Cardiomyopathy
* Gastrointestinal disorders particularly those associated with a high risk of perforation or fistula formation including:

  * Any of the following that have not resolved within 28 days before the first dose of study treatment

    * Intra-abdominal tumor/metastases invading GI mucosa
    * Active peptic ulcer disease
    * Diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis
    * Malabsorption syndrome
  * Any of the following within 6 months before the first dose of study treatment:

    * Abdominal fistula
    * Gastrointestinal perforation
    * Bowel obstruction or gastric outlet obstruction
    * Intra-abdominal abscess; Note: complete resolution of an intra-abdominal abscess must be confirmed prior to initiating treatment with cabozantinib even if the abscess occurred more than 6 months before the first dose of study treatment
* Other disorders associated with a high risk of fistula formation including percutaneous endoscopic gastrostomy (PEG) tube placement within 3 months before the first dose of study therapy
* Other clinically significant disorders such as:

  * Severe active infection requiring systemic treatment within 14 days before the first dose of study treatment
  * Serious non-healing wound/ulcer/bone fracture within 28 days before the first dose of study treatment
  * History of organ transplant
  * Concurrent uncompensated hypothyroidism or thyroid dysfunction within 7 days before the first dose of study treatment (for asymptomatic patients with an elevated thyroid stimulating hormone [TSH], thyroid replacement may be initiated if clinically indicated without delaying the start of study treatment)
  * History of major surgery as follows:

    * Major surgery within 3 months of the first dose of cabozantinib; however, if there were no wound healing complications, patients with rapidly growing aggressive cancers, may start as soon as 6 weeks if wound has completely healed post-surgery
    * Minor surgery within 1 month of the first dose of cabozantinib if there were no wound healing complications or within 3 months of the first dose of cabozantinib if there were wound complications excluding core biopsies and Mediport placement
  * In addition, complete wound healing from prior surgery must be confirmed at least 28 days before the first dose of cabozantinib irrespective of the time from surgery
* The subject is unable to swallow tablets
* History of severe hypersensitivity reaction to any monoclonal antibody
* The subject is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee
* For disease specific studies: the subject has had evidence within 2 years of the start of study treatment of another malignancy which required systemic treatment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cabozantinib, nivolumab, ipilimumab or other agents used in study
* Pregnant women are excluded from this study because cabozantinib is a tyrosine kinase inhibitor with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with cabozantinib, breastfeeding should be discontinued if the mother is treated with cabozantinib; these potential risks may also apply to other agents used in this study
* Human immunodeficiency virus (HIV)-positive patients are eligible if on stable dose of highly active antiretroviral therapy (HAART), CD4 counts are greater than 350 and viral load is undetectable
* Patients are excluded if they have a positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids, should be excluded; these include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease; patients with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible; patients with rheumatoid arthritis and other arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible
* Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event)
* Patients are excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration; inhaled or topical steroids and adrenal replacement doses < 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease; patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption); physiologic replacement doses of systemic corticosteroids are permitted, even if < 10 mg/day prednisone equivalents; a brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted
* Patients who have had evidence of active or acute diverticulitis, intra-abdominal abscess, GI obstruction and abdominal carcinomatosis which are known risk factors for bowel perforation should be evaluated for the potential need for additional treatment before coming on study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2015-07-22 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Recommended phase II dose (Phase I) | Up to 4-6 weeks
  Will be defined as the highest dose for which no more than 1/6 patients experience a dose limiting toxicity evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. The safe dose level of cabozantinib and nivolumab, as well as of cabozantinib, nivolumab, and ipilimumab will be established.
Incidence of adverse events (Phase I) | Up to 30 days post treatment
  Will be evaluated according National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. The safety and tolerability of a novel dose of cabozantinib, nivolumab and ipilimumab in patients with genitourinary cancer will be assessed.

SECONDARY OUTCOMES:
Clinical response rate | Up to 3 years
  Will be assessed by Response Evaluation Criteria in Solid Tumors 1.1 and Immune-Related Response Criteria. The response rate may be used to guide the further development of the combinations.
Fraction of patients who have been identified as being alive and progression free at two months | At 2 months
  May be determined as well and reported on both arms. This fraction will be considered as a secondary endpoint for the expansion cohorts as well, and this information may be used to guide the further development of the combinations. A Kaplan-Meier curve for progression free survival will also be presented as a secondary endpoint, in addition to reporting the fraction without progression at two months.
PDL-1 and MET expression | Up to day 1 of final cycle
  PDL-1 and MET expression data will be obtained in patients with urothelial carcinoma checkpoint inhibition naive, clear cell renal cell carcinoma, adenocarcinoma of the bladder, squamous cell carcinoma of the bladder, urothelial carcinoma with prior checkpoint inhibition therapy, and penile cancer. Data will be obtained in pre- and post-treatment biopsies and analyze, in at least an exploratory fashion, their association to response or clinical benefit.

OTHER OUTCOMES:
Overall response rate in patients receiving ipilimumab challenge/re-challenge | Up to 3 years
  The overall response rates determined at this time point will be combined and reported along with 95% confidence intervals.
Progression free survival in bone-only urothelial carcinoma | Up to 3 years
  Patients with bone-only disease will be enrolled and evaluated using progression free survival for a descriptive analysis of the effect of treatment. In addition, if PDL-1 or MET data are obtained in this small cohort, exploratory and descriptive analyses may be done as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea B Apolo, Principal Investigator — National Cancer Institute LAO
Locations (8):
- United States (8):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - NCI - Center for Cancer Research, Bethesda, Maryland
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

REFERENCES:
- [Derived] Apolo AB, Girardi DM, Niglio SA, Nadal R, Kydd AR, Simon N, Ley L, Cordes LM, Chandran E, Steinberg SM, Lee S, Lee MJ, Rastogi S, Sato N, Cao L, Banday AR, Boudjadi S, Merino MJ, Toubaji A, Akbulut D, Redd B, Bagheri H, Costello R, Gurram S, Agarwal PK, Chalfin HJ, Valera V, Streicher H, Wright JJ, Sharon E, Figg WD, Parnes HL, Gulley JL, Saraiya B, Pal SK, Quinn D, Stein MN, Lara PN, Bottaro DP, Mortazavi A. Final Results From a Phase I Trial and Expansion Cohorts of Cabozantinib and Nivolumab Alone or With Ipilimumab for Advanced/Metastatic Genitourinary Tumors. J Clin Oncol. 2024 Sep 1;42(25):3033-3046. doi: 10.1200/JCO.23.02233. Epub 2024 Jul 2. PMID 38954785
- [Derived] Girardi DM, Niglio SA, Mortazavi A, Nadal R, Lara P, Pal SK, Saraiya B, Cordes L, Ley L, Ortiz OS, Cadena J, Diaz C, Bagheri H, Redd B, Steinberg SM, Costello R, Chan KS, Lee MJ, Lee S, Yu Y, Gurram S, Chalfin HJ, Valera V, Figg WD, Merino M, Toubaji A, Streicher H, Wright JJ, Sharon E, Parnes HL, Ning YM, Bottaro DP, Cao L, Trepel JB, Apolo AB. Cabozantinib plus Nivolumab Phase I Expansion Study in Patients with Metastatic Urothelial Carcinoma Refractory to Immune Checkpoint Inhibitor Therapy. Clin Cancer Res. 2022 Apr 1;28(7):1353-1362. doi: 10.1158/1078-0432.CCR-21-3726. PMID 35031545
- [Derived] Apolo AB, Nadal R, Girardi DM, Niglio SA, Ley L, Cordes LM, Steinberg SM, Sierra Ortiz O, Cadena J, Diaz C, Mallek M, Davarpanah NN, Costello R, Trepel JB, Lee MJ, Merino MJ, Bagheri MH, Monk P, Figg WD, Gulley JL, Agarwal PK, Valera V, Chalfin HJ, Jones J, Streicher H, Wright JJ, Ning YM, Parnes HL, Dahut WL, Bottaro DP, Lara PN Jr, Saraiya B, Pal SK, Stein MN, Mortazavi A. Phase I Study of Cabozantinib and Nivolumab Alone or With Ipilimumab for Advanced or Metastatic Urothelial Carcinoma and Other Genitourinary Tumors. J Clin Oncol. 2020 Nov 1;38(31):3672-3684. doi: 10.1200/JCO.20.01652. Epub 2020 Sep 11. PMID 32915679